CLINICAL TRIAL: NCT05048823
Title: Osteopathic Bowel Techniques and Their Effects on the Autonomic Nervous and Pain Pressure Sensitivity: Randomized Clinical Trial
Brief Title: Osteopathic Bowel Techniques and Their Effects on the Autonomic Nervous System in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Docusse de Osteopatia e Terapia Manual (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17249119.2.0000.5515
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Volunteers will be randomly distributed into two groups called intervention protocol and placebo protocol. Only the participant and the outcome assessor will be blinded to the protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Protocol (Experimental): Visceral techniques for the gastrointestinal system
  Interventions: Other: Visceral Osteopathic Techniques
- Placebo Protocol (Sham Comparator): simulated visceral techniques in the region of the gastrointestinal system, without therapeutic intent
  Interventions: Other: Simulated visceral techniques

INTERVENTIONS:
Other: Visceral Osteopathic Techniques — Generalized Discharge Technique of the Peritoneum and Intestinal Wings, Mobilization of the Cecum, Technique for the Root of the Mesentery, Release of the D1-D2 Angle, Technique for the Sigmoid Colon
  Arms: Intervention Protocol
Other: Simulated visceral techniques — Simulated visceral techniques in the region of the gastrointestinal system
  Arms: Placebo Protocol

SUMMARY:
INTRODUCTION: The autonomic nervous system (ANS) is responsible for controlling several visceral functions, including the motility and secretion of the gastrointestinal system (GIS). Alterations in the functioning of the ANS can directly influence the physiological mechanisms of the GIS. Due to the importance of the ANS in the control of various body functions, strategies aimed at acting in this system have become extremely important and have been widely used in the literature. Some of the studies involving ANS analysis have shown that osteopathic manipulative treatment is able to promote a reduction in sympathetic ANS activity and an increase in parasympathetic ANS activity in asymptomatic youngsters, however, none of them addressed the GIS, already known to be influenced by autonomic fibers. OBJECTIVE: To evaluate the immediate effects of GIS-directed osteopathic techniques on ANS behavior and pain sensitivity to pressure in young people without symptoms of gastrointestinal disorders. METHODS: The present study is characterized by a randomized, single-blind clinical trial, in which 42 asymptomatic individuals will be recruited, regardless of gender, aged between 18 and 30 years. Volunteers will be randomly distributed into two groups called intervention protocol and placebo protocol. The intervention protocol will be performed by a professional with 10 years of clinical experience in the field of Osteopathy and will perform the techniques of Generalized Discharge of the peritoneum and intestinal wings, Mobilization of the Cecum, technique for the Mesentery Root, Release of the D1-D2 angle, technique for the Sigmoid Colon. The approximate duration of the set of techniques will be 15 minutes with the volunteers positioned supine on a stretcher. The placebo protocol will apply in the same way regarding the positioning and duration of the techniques. The therapist will position the hands in the same regions of the intervention protocol, maintaining superficial contact for 3 minutes in each region, without therapeutic intent. Volunteers will be evaluated for outcomes before and immediately after performing the protocols. The heart rate variability will be measured by capturing the intervals between each beat in ms, using a heart rate monitor and extracting the linear indices in the domain of time, frequency and geometric heart rate variability. The pressure pain threshold will also be measured using a pressure algometer that will be positioned in the vertebral region of T5-L3. Comparisons of variables (indices of HRV and pressure pain threshold) between the intervention protocol group and placebo protocol will be performed using the Student's T test (normal data) or the Mann-Whitney test (non-normal data). All results will be discussed at the 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

-Health individuals

Exclusion Criteria:

* Participants with neurological impairment and/or pathologies that interfere with autonomic behavior
* smokers
* diagnosis of pulmonary disease
* Participants with theoretical and/or practical knowledge about the techniques that will be applied in the protocol

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | Immediately after intervention
  The HRV data will be analyzed using linear methods, analyzed in the time and frequency domains and using geometric indices.

SECONDARY OUTCOMES:
Pressure pain threshold | Immediately after intervention
  Pressure pain threshold will be assessed using a mechanical device (algometer), known to quantify pain intensity at a specific point through local pressure. The pain threshold will be considered through the minimum pressure necessary to induce pain in the assessed region. The points evaluated in this study correspond to the thoracic and lumbar levels of T5-L3

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Kastelianne, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Will be shared with other researchers when requested
Supporting Information: Study Protocol, SAP
Time Frame: After one year from publication
Access Criteria: To request the data, please contact nupi@idot.com.br